CLINICAL TRIAL: NCT05983016
Title: Automated Three-dimensional Ultrasound Bridges the Gap Between Novices and Experts in Diameter Assessment of Abdominal Aortic Aneurysms
Brief Title: Automatic Abdominal Aortic Aneurysm Diameter Measurement
Status: Completed | Type: Observational
Sponsor: Natasha Monzon Svendsen (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor-Investigator, Natasha Monzon Svendsen, MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-20001116
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: AAA - Abdominal Aortic Aneurysm
Keywords: Ultrasound; Three dimensional ultrasound; Abdominal aortic aneurysm; Sonography; 3D ultrasound
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients: All ten patients had their abdominal aortic aneurysm measured by experts and novices using both two-dimensional and three-dimensional ultrasound
  Interventions: Device: Philips EPIQ-7, Philips Healthcare, Bothell, WA, USA

INTERVENTIONS:
Device: Philips EPIQ-7, Philips Healthcare, Bothell, WA, USA — All patients had their abdominal aortic aneurysm maximum anterior-posterior diameter estimated with two-dimensional ultrasound using a 5 MHz curved array transducer (Philips® C5-1 transducer, Philips Healthcare, Bothell, WA, USA).
  After the acquisition, a three-dimensional ultrasound acquisition was performed with a 3D-matrix transducer (Philips® X6-1 transducers, Philips Healthcare, Bothell, WA, USA).

SUMMARY:
Managing abdominal aortic aneurysms currently relies on diameter assessment with ultrasound. Diameter reproducibility with two-dimensional ultrasound is challenging, and requires experienced operators. A novel automatic three-dimensional ultrasound system has the potential to facilitate more precise diameter measurements than two-dimensional ultrasound. This study aimed to assess the variance of abdominal aortic aneurysm diameter measurements among ultrasound novices and experts by comparing two-dimensional ultrasound with the three-dimensional ultrasound system in a clinical setting.

Ten patients under abdominal aortic aneurysm surveillance were examined by 29 ultrasound-operators: 13 experts and 16 novices. The experts were sonographers and physicians highly experienced in abdominal aortic aneurysm ultrasound, and the novices were medical students and junior residents with sparse ultrasound experience.

ELIGIBILITY:
Inclusion Criteria:

-Patients with an abdominal aortic aneurysm > 3 cm.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The ten patients were selected from a large vascular surgery outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Abdominal aortic aneurysm measurement variance between novices and experts | One week
  The primary outcome was to test the variance of abdominal aortic aneurysm diameter measurements by comparing expert and novice ultrasound operators using conventional 2D-ultrasound and 3D-software assisted ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Vascular Surgery, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided